CLINICAL TRIAL: NCT04791462
Title: Observational Descriptive Study of Stress Symptoms Related to the COVID-19 Outbreak in a Cohort of Osteoarthritis Patients
Brief Title: COVID-19 in Osteoarthritis Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0109
Record Dates: First submitted 2021-02-26; First posted 2021-03-10 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Osteoarthritis
Keywords: lower limbs; anxiety; stress; Covid19
MeSH Terms: conditions — Osteoarthritis; Anxiety Disorders; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — NC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
While the coronavirus pandemic has spread rapidly around the world, it has generated a considerable degree of fear, concern and anxiety among the population in general and among certain groups in particular, such as older persons. Initial findings from studies in China indicated the presence of moderate to severe psychological impact in a significant proportion of individuals and an increased prevalence of post-traumatic stress symptoms. It should also be noted that other types of symptoms, such as anxiety and depression, appeared to persist over time and to a greater extent.

Osteoarthritis can develop in any joint, but most often affects the knees, hands and hips. People with osteoarthritis are often older and sometimes more frail than the general population. The main recommendations for non-drug treatment of osteoarthritis include education, physical activity and structured exercise programmes with or without weight reduction. Due to the confinement associated with COVID-19, many patients have had to stop exercise/physical activity and postpone prosthetic surgery. Apart from the context of delay in surgery, there is little data available on the impact of the pandemic on people with arthritis. Several questions are therefore still pending concerning the impact of the pandemic on these patients.

The investigators hypothesise that the following therapeutic modalities have been disrupted during this period: access to care, scheduling of prosthetic surgery, consumption of painkillers or NSAIDs, recourse to physical activities, recourse to physiotherapy sessions, weight changes, level of pain.... Our objective is to evaluate the physical, social, psychological and behavioural consequences of the COVID-19 pandemic in a cohort of osteoarthritis patients.

ELIGIBILITY:
Inclusion criteria:

- OA patients

Exclusion criteria:

* active or passive opposition of the patient and / or its legal representatives to participate in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a physician-confirmed diagnosis of osteoarthritis of the lower limbs
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Assessing the state of post-traumatic stress | 12 months
  Assessing the state of post-traumatic stress in OA patients 12 months after the start of the COVID-19 outbreak (use of the PCL-5 score, with a discriminating threshold score of 38 out of a total score of 80)

SECONDARY OUTCOMES:
To evaluate the level of anxiety/depression | 1 day
  To evaluate the level of anxiety/depression in the OA patient defined by the HAD score.
  HAD score: Hospital Anxiety and Depression score: Higher values means poor outcome, min 0, max 42
To evaluate the level of stress perceived | 1 day
  To evaluate the level of stress perceived by the OA patient as defined by the PSS14 score.
  PSS14 score: Perceived Stress Scale , 14 questions, Rating (0 = Never, 1 = Almost never, 2 = Sometimes, 3 = Quite often, 4 = Very often): Higher score = poor outcome 3/ PCL-5: Post-Traumatic Stress Disorder Checklist Scale, version DSM-V, Items are rated from 0 "not at all" to 4 "extremely". 20 questions, Higher score = poor outcome PCL-5: Post-Traumatic Stress Disorder Checklist Scale, version DSM-V, Items are rated from 0 "not at all" to 4 "extremely". 20 questions, Higher score = poor outcome
To evaluate the level of physical activity | 1 day
  To evaluate the level of physical activity in the OA patient defined by the IPAQ score.
  IPAQ: International Physical Activity Questionnaire - Craig et al. 2003; Short version (7 questions). The questionnaire classifies the subject according to 3 levels of activity: inactive, moderate, high
Assess demographic influencing perceived stress, anxiety/depression, physical activity, post-traumatic stress disorder | 1 day
  Assess demographic influencing perceived stress, anxiety/depression, physical activity, post-traumatic stress disorder

CONTACTS AND LOCATIONS:
Overall Officials: Yves-Marie PERS, M.D., Ph. D., Principal Investigator — UH Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC